CLINICAL TRIAL: NCT04168320
Title: CLINICAL EXPLORATION OF THE NON-TARGETED EFFECTS OF STEREOTACTIC RADIOTHERAPY IN PATIENTS WITH UNRESECTABLE BULKY TUMORS TREATED BY PARTIAL HIGH-DOSE IRRADIATION OF HYPOXIC TUMOR SEGMENT: PHASE I PROOF OF PRINCIPLE TRIAL.
Brief Title: SBRT-based PArtial Tumor Irradiation of HYpoxic Segment
Acronym: SBRT-PATHY
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because of the prolonged/poor patient recruitment
Sponsor: Klinikum Klagenfurt am Wörthersee (Other)
Responsible Party: Principal Investigator, Slavisa Tubin, Vice-Chairman of the Radiation Oncology Institute, Klinikum Klagenfurt am Wörthersee, Klinikum Klagenfurt am Wörthersee
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A21/18
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Bystander Effect; Abscopal Effect; Unresectable Malignant Solid Neoplasm; Bulky Tumors
Keywords: Phase I; Bystander effect; Abscopal effect; Tumor hypoxia

STUDY DESIGN:
Intervention Model Description: Starting two weeks prior to the initiation of radiotherapy serial, 7x blood samples will be taken every two days, excluding the weekend (for example, if starting on a Monday: Monday-Wednesday-Friday-Monday-Wednesday-Friday and Monday), but also on the day of the first radiotherapy treatment, to define the serial high-sensitivity C-reactive protein (hs-CRP) test, LDH and white cell differential count (leucocytes: neutrophils, basophils, eosinophils, lymphocytes, monocytes).
  Data from the assays will be assembled in a spreadsheet and analyzed for levels and cyclical fluctuations to determine each patient's idiosyncratic immune cycle's periodicity and then each patient's time-position of initiation of treatment and response to therapy. Radiotherapy will be administered to the arm 1 (13 patients) at an estimated "less favorable time-position", while it will be administered to the arm 2 (13 patients) at an estimated "most favorable time-position in immune cycle".
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Less favorable time-position in immune cycle (Active Comparator): Starting two weeks prior to the initiation of radiotherapy serial, 7x blood samples will be taken every two days, excluding the weekend (for example, if starting on a Monday: Monday-Wednesday-Friday-Monday-Wednesday-Friday and Monday), but also on the day of the first radiotherapy treatment, to define the serial high-sensitivity C-reactive protein (hs-CRP) test, LDH and white cell differential count (leucocytes: neutrophils, basophils, eosinophils, lymphocytes, monocytes). Data from the assays will be assembled in a spreadsheet and analyzed for levels and cyclical fluctuations to determine each patient's idiosyncratic immune cycle's periodicity and then each patient's time-position of initiation of treatment and response to therapy.
  SBRT-PATHY will be administered to this arm at an estimated "less favorable time-Position in immune cycle".
  Interventions: Radiation: SBRT-PATHY (SBRT-based PArtial Tumor irradiation targeting HYpoxic segment)
- Most favorable time-position in immune cycle (Experimental): Starting two weeks prior to the initiation of radiotherapy serial, 7x blood samples will be taken every two days, excluding the weekend (for example, if starting on a Monday: Monday-Wednesday-Friday-Monday-Wednesday-Friday and Monday), but also on the day of the first radiotherapy treatment, to define the serial high-sensitivity C-reactive protein (hs-CRP) test, LDH and white cell differential count (leucocytes: neutrophils, basophils, eosinophils, lymphocytes, monocytes). Data from the assays will be assembled in a spreadsheet and analyzed for levels and cyclical fluctuations to determine each patient's idiosyncratic immune cycle's periodicity and then each patient's time-position of initiation of treatment and response to therapy.
  SBRT-PATHY will be administered to this arm at an estimated "most favorable time-position in immune cycle".
  Interventions: Radiation: SBRT-PATHY (SBRT-based PArtial Tumor irradiation targeting HYpoxic segment)

INTERVENTIONS:
Radiation: SBRT-PATHY (SBRT-based PArtial Tumor irradiation targeting HYpoxic segment) — Novel stereotactic high-dose partial irradiation of the hypoxic segment of bulky tumors.

SUMMARY:
This study uses an unconventional radiotherapy schedule developed at our institute, consisting of a short course high-dose partial irradiation targeting exclusively the hypoxic segment of a bulky tumors, which in our preliminary study has shown to be capable of inducing abscopal and bystander effects. This approach is delivered by using a stereotactic radiotherapy technique so as to spare nearby organs at risk including the peritumoral immune microenvironment from irradiation as much as possible. Our approach consists of a single or up to 3 radiotherapy doses of at least 10 Gy per fraction prescribed to the 70% isodose line encompassing the hypoxic target volume. Radiotherapy will be administered at the precise timing determined specifically for each patient based on the serially mapped homeostatic immune fluctuations by monitoring the blood levels of the cytokines and inflammatory markers over the 2 weeks prior to irradiation. This is done in order to synchronize the radiation treatment with the favorable, most active anti-tumor immune system phase, so as to stimulate and increase anti-tumor immune system activity.

This is a monocentric, prospective, two-arm, phase I proof of principle study in which the investigator will enroll subjects with oligometastatic and/or locally advanced (N+) cancers with at least one "bulky" lesion (maximum diameter of at least 6 cm or greater). Patients with life expectancy of at least 3 months, who are ineligible for systemic therapy or experience disease progression with systemic therapies will be included. Radiotherapy will be administered to arm 1 at an estimated "less favorable time-position in immune cycle", while the second arm will have it administered at the estimated "most favorable time-position in immune cycle".

The primary endpoint will be the response rate of the non-targeted effects both bystander (local, at the level of the partially treated bulky tumor) and abscopal (distant, at the non-treated metastatic sites), defined as a tumor regression of at least 30%. Secondary endpoints will be safety, survival and analysis of the best timing for the administration of radiotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of our new method for high dose partial irradiation of the hypoxic tumor segment of bulky masses in terms of the intentional induction of the non-targeted effects of radiotherapy in patients with metastatic or locally advanced (N+) malignancies who are ineligible for, or currently in progression under systemic therapies. By mapping the homeostatic immune fluctuations serially, and by monitoring the blood levels of the cytokines and inflammatory markers over the 2 weeks prior to irradiation, radiotherapy will be administered at the precise, optimal timing in order to stimulate and to increase anti-tumor immune system activity.

Primary endpoint: bystander (local) and abscopal (distant, metastatic or lymph nodal sites) response rates.

Secondary endpoints: overall safety and tolerability profile of our new radiotherapy method, progression-free survival rates at local and distant sites, as well as overall survival rates, efficacy of this regimen in palliating symptoms, neoadjuvant potential of this novel radiotherapy for unresectable/borderline resectable bulky lesions, optimal timing for radiotherapy to be administered based on the fluctuating/oscillating suppressed anti-tumor immune response.

This monocentric, two-arm prospective phase I proof of principle trial will enroll 26 patients from a single institution: KABEG Klinikum Klagenfurt am Woerthersee, Austria.

During the visit, and after clinical examination, patients will be eligible if they satisfy the inclusion criteria for participation in this pilot study on the use of the novel stereotactic radiotherapy technique which will consist of partial irradiation of exclusively hypoxic segments of their bulky tumors, with 1-3 high dose fractions of radiotherapy based on the tumor's site, volume and its relationship with nearby organs. The irradiation will take place within 3 weeks of clinical examination. After the treatment, the patient will be regularly followed for the evaluation of all endpoints. If any severe toxicity (grade ≥3 per CTCAE v 4.3 criteria) occurs in the first 7 evaluable patients, the trial will stop. Safety reviews will continue on an ongoing basis, provided that severe toxicities do not occur in more than 15% of patients. In the case of eventual disease progression during the follow-up, the patients will be offered additional local (radiotherapy) or systemic (chemotherapy, immunotherapy, hormonal therapy) treatment if indicated by current NCCN (National Comprehensive Cancer Network) treatment recommendations and guidelines.

Routine surveillance computerized axial tomography (CT) imaging of the whole body will be performed beginning at 1 month (+/- 3 days) after treatment to allow for endpoint assessment - or before in any case of clinical suspicion of disease progression. Routine CT imaging surveillance will continue per standard of care. Patients will also be followed clinically with physical and laboratory examinations as indicated.

Tumor assessments will be completed on the CRF using RECIST v1.1. criteria. Radiographic and clinical evaluations will be conducted with the same schedule. The investigator will assess anti-tumor activity based on radiological assessments and clinical evaluations of patients using RECIST v1.1 at baseline, 1 and 2 months post-treatment, and every 3 months thereafter until confirmed disease progression per RECIST v1.1, regardless of the discontinuation of study treatment or the initiation of subsequent anti-cancer therapy. Radiological tumor assessments will also be conducted whenever disease progression is suspected (e.g. symptomatic deterioration or physical examination findings suggestive of mucosal recurrence).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic biopsy proven malignant cancer with at least one "bulky" (diameter of at least 6 cm or greater) lesion, or in the case of a biopsy missing for any reason-progression of the suspicious lesion evaluated on at least 2 consecutive radiological examinations,
* Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluation,
* Ineligibility for systemic therapy or being in progression under systemic therapy,
* A minimum time interval of four weeks from the last dose of systemic therapy before radiotherapy,
* Median life expectancy of >3 months,
* Age > 18 years at the time of study entry,
* Adequate bone marrow function: Haemoglobin ≥ 9.0 g/dL, absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3), platelet count ≥ 100 x 109/L (>100,000 per mm3),
* Female subjects must either be of non-reproductive potential (i.e. post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry,
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.

Exclusion Criteria:

* Patients without metastatic cancer (regional metastatic lymph nodes considered as metastatic),
* Patients without bulky lesions,
* Median life expectancy of less than three months,
* Patients with prior radiation therapy to the same site,
* Contraindication to IV iodine contrast medium administration, particularly estimated glomerular filtration rate (GFR) less than 45 mL/min/1.73 m2,
* History of autoimmune disease,
* Current or prior use of immunosuppressive medication within 28 days before enrollment with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid,
* History of primary immunodeficiency,
* History of allogeneic organ transplant,
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent,
* Known history of previous clinical diagnosis of tuberculosis,
* History of leptomeningeal carcinomatosis,
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control,
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results,
* Subjects with uncontrolled seizures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Bystander and abscopal effects | 6 months
  Rates of significant (30% or more) tumor regression at the level of both the partially treated bulky tumors (bystander effects) and unirradiated oligometastases and/or regional lymph nodes (abscopal effect).

SECONDARY OUTCOMES:
Overall survival | Up to 100 weeks
  The length of time from the start of treatment for a cancer, that patients diagnosed with the disease are still alive.
Progression-free survival | Up to 100 weeks
  The length of time during and after the treatment of a cancer, that a patient lives without disease-progression.
Patient-reported outcome (PRO) | 3 months
  Health outcome directly reported by the patient who experienced the cancer-related symptoms.
Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 100 weeks
  Clinician reported radiation related toxicity as a standardized system to quantify or grade the severity of adverse events that occur during or after radiation treatment.
Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 6 months
  The assessments of tumor response to radiotherapy will be performed using RECIST v1.1. criteria at 1 and 2 months post-treatment, and every 3 months thereafter using CT, MRI or PET-CT to assess the neoadjuvant potential of SBRT-PATHY expressed as significant (>30% tumor-volume reduction in respect to initial tumor volume) downsizing of unresectable bulky tumors into resectable tumors.
Timing | 6 months
  Determination of the optimal timing for radiotherapy treatment to be administered by correlating the clinical outcomes with the phase or position on the immune cycle at which the treatment occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Slavisa Tubin, M.D., Principal Investigator — KABEG Klinikum Klagenfurt
Locations (1):
- KABEG Klinikum Klagenfurt, Institute for Radiation Oncology, Klagenfurt, Carinthia, Austria